CLINICAL TRIAL: NCT05433090
Title: An Inpatient Advance Care Planning Intervention for Older Patients With Hematologic Malignancies
Acronym: Inpatient SICP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UOCPC22039
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancies
Keywords: Advance Care Planning Intervention; Serious Illness Conversation; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention used in this study is an inpatient advance care planning intervention. We will adapt the Serious Illness Care Program, an evidence-based intervention that promotes serious illness conversation between patients and clinicians, to be used by advance practice providers and hematology/oncology fellow physicians in the inpatient setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients will participate in an inpatient advance care planning intervention.
  Interventions: Behavioral: Inpatient serious illness care program

INTERVENTIONS:
Behavioral: Inpatient serious illness care program — Inpatient advance care planning intervention that will be delivered by advanced care practitioners or hematology/oncology fellow physicians. The intervention will be an adapted version of the serious illness care program.

SUMMARY:
This is a pilot study to assess the preliminary efficacy of an inpatient advance care planning intervention on outcomes in older patients with hematologic malignancies

DETAILED DESCRIPTION:
Older adults with hematologic malignancies receive more aggressive inpatient care at the end of life compared to patients with solid tumors. Advance care planning may promote early serious illness conversations for patients with hematologic malignancies, leading to less aggressive healthcare utilization at the end of life. This pilot aims to assess the preliminary efficacy of an inpatient advance care planning intervention on outcomes in older patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* A diagnosis of hematologic malignancy [including but not limited to acute leukemia, myeloid malignancies (e.g., atypical CML, MDS/MPN overlap syndromes, CMML), multiple myeloma, lymphoma, or any other hematologic malignancies based on the primary oncologist's judgment]
* Able to provide informed consent
* Being managed in the inpatient setting
* English-speaking

Exclusion Criteria:

• None

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A final study protocol including a description of the study participants, measurements, data, and analyses will be available on clinicaltrials.gov before the results are published.
Supporting Information: Study Protocol
Time Frame: Data will be available for 7 years after the study closes, from approximately November 15, 2025 until November 15, 2030.
Access Criteria: The protocol is publicly available on ClinicalTrials.gov.

REFERENCES:
- [Background] LoCastro M, Baran AM, Liesveld JL, Huselton E, Becker MW, O'Dwyer KM, Aljitawi OS, Baumgart M, Snyder E, Kluger B, Loh KP, Mendler JH. Portable medical orders and end-of-life measures in acute myeloid leukemia and myelodysplastic syndromes. Blood Adv. 2021 Dec 28;5(24):5554-5564. doi: 10.1182/bloodadvances.2021004775. PMID 34525170
- [Result] Marissa Locastro, Ying Wang, Soroush Mortaz-Hedjri, Danielle Frumusa, Tracy Natale, Jessica Cohen, Nicole Yates, Jenna Podlucky, Tristan Yu, Thomas Carroll, Jane L. Liesveld, Megan Baumgart, Sandra Sabtka, Dwight Hettler, Nicole Kaplan, Jason H. Mendler, Kah Poh Loh; An Inpatient Advance Care Planning Intervention for Older Patients with Hematologic Malignancies: A Single-Arm Pilot Study. Blood 2024; 144 (Supplement 1): 5054. doi: https://doi.org/10.1182/blood-2024-206137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients being managed in the inpatient setting at the University of Rochester Medical Center (URMC) Wilmot Cancer Institute (WCI), were identified by treating physicians, APPs, hematology/oncology fellows, nurses, and study coordinators. Patients were recruited from November 2022 to October 2024.
Pre-assignment Details: 57 patients were approached, and 41 consented (consent rate: 71.9%). The most common reasons patients declined to participate were a reluctance to complete surveys (n=8), feeling overwhelmed by their current situation (n=5), or a belief that discussing their preferences with the care team would not be helpful (n=3).
Groups:
- Advanced Care Planning: This is a single-arm pilot study. After completing baseline measures, all patients received an inpatient Advanced Care Planning (ACP) intervention. Before the visit, patients received a preparation pamphlet. The APP/hematology/oncology fellow used the "Serious Illness Care Guide" during the ACP intervention to discuss advanced care planning and end of life care with the patient. At the end of the visit, patients received a "Family Guide" to help communicate with their family about the visit.
Period: Overall Study
Arm/Group | Advanced Care Planning
Started | 41
Completed ACP Intervention | 38
Completed | 35
Not Completed | 6
Not completed — Patient Discharged Before ACP Intervention | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: All participants who completed baseline measures (n = 41).
Arm/Group | Advanced Care Planning
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Education [Count of Participants; unit: Participants] — Patient response to: "Highest level of education achieved."
  Participants
    High school or below | 12
    Training after high school or some college/university | 12
    College/University graduate | 11
    Post Graduate level | 5
    Other | 1
Marital status [Count of Participants; unit: Participants] — Patient response to: "Marital status."
  Participants
    Married/long term, committed significant other | 24
    Divorced | 3
    Single | 5
    Widowed | 9
Employment status [Count of Participants; unit: Participants] — Patient response to: "Employment status."
  Participants
    Employed | 10
    Retired | 28
    Unemployed | 1
    Homemaker | 0
    Other | 2
Caregiver living with the patient [Count of Participants; unit: Participants] — Patient response to: "Who do you live with?"
  Participants
    Partner (spouse/significant other) | 25
    Child/children | 1
    None | 15
Caregiver not living with the patient [Count of Participants; unit: Participants] — Patient response to: "Do you have a caregiver who is not living with you?"
  Participants
    Partner (spouse/significant other) | 5
    Child/children | 8
    Other relative(s) | 2
    None | 26
Cancer diagnosis [Count of Participants; unit: Participants]
  Acute lymphoblastic leukemia | 3
  Acute myeloid leukemia | 25
  Central Nervous System Lymphoma | 1
  Lymphoma | 3
  Multiple myeloma | 4
  Myelodysplastic syndrome | 4
  Plasma cell leukemia | 1
Cancer diagnosis duration [Count of Participants; unit: Participants] — The length of time between date of diagnosis and baseline date.
  Participants
    <6 months | 24
    >= 6 months | 17
Cancer health literacy [Count of Participants; unit: Participants] — Cancer Health Literacy Test-6 (CHLT-6) was used to assess patient cancer health literacy.
  Participants
    Adequate literacy | 39
    Limited literacy | 2

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate
Description: Retention rate is the percentage of consented patients who completed the ACP intervention visit. A retention rate of >70% was considered feasible.
Time Frame: From consent until completion of the ACP intervention visit, usually within 1 week.
Population: All consented participants who underwent baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Care Planning
Number analyzed (Participants) | 41
Participants
  Retained - completed ACP intervention | 38
  Not retained - didn't complete ACP intervention | 3

2. Secondary Outcome: Advance Directive Completion - HCP
Description: Data on the patient's completion of scanned healthcare proxy form that was completed with their physician was collected via the electronic medical record. This is expressed as a percentage.
Time Frame: From baseline (pre-intervention) to 1 year post-intervention. The time interval is approximately 1 year.
Population: All participants who consented and completed baseline measures. Baseline and post-intervention data represent paired data from the same participants who completed both timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Care Planning
Number analyzed (Participants) | 41
Participants
  Baseline: HCP Completed | 23
  Baseline: HCP Not Completed | 18
  After ACP Intervention: HCP Completed | 31
  After ACP Intervention: HCP Not Completed | 10

3. Secondary Outcome: Advance Directive Completion - MOLST
Description: Data on the patient's completion of scanned medical order for life sustaining treatment (MOLST) form that was completed with their clinician was collected via the electronic medical record. This is expressed as a percentage.
Time Frame: From baseline (pre-intervention) to 1 year post-intervention. The time interval is approximately 1 year.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Care Planning
Number analyzed (Participants) | 41
Participants
  Baseline: MOLST Completed | 7
  Baseline: MOLST Not Completed | 34
  After ACP Intervention: MOLST Completed | 20
  After ACP Intervention: MOLST Not Completed | 21

ADVERSE EVENTS:
Time Frame: Patient adverse events and mortality were collected and reported from enrollment until the end of follow-up, up to approximately 2 months after enrollment.
Arm/Group | Advanced Care Planning
All-Cause Mortality (participants affected / at risk) | 2/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

LIMITATIONS AND CAVEATS:
This was a single-center study with a relatively small sample size (enrolled n=41).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05433090/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT05433090/ICF_001.pdf